## PROTOCOL

Effect of Postoperative Oral Carbohydrate Administration in Total Keen Arthroplasty
Patients
October 16,2022

# Effect of Postoperative Oral Carbohydrate Administration in Total Keen Arthroplasty

#### 1. Research background

In recent years, the concept of accelerated rehabilitation surgery (enhanced recovery after surgery, ERAS) has developed vigorously, using a series of optimized evidence-based medical support with preoperative, intraoperative and postoperative programs to reduce postoperative physiological and psychological stress trauma response, so as to achieve the goal of accelerating patient rehabilitation<sup>[1]</sup>. Perioperative fasting water ban management is an important component of ERAS. Studies have found that prolonged preoperative drinking and fasting will increase the postoperative insulin resistance, cause hypertension, and increase the risk of postoperative infection, which is not conducive to the postoperative recovery of [2]. Oral carbohydrates for at least 2h before anesthesia can reduce the perioperative stress response, improve patient comfort and satisfaction, and promote the postoperative rehabilitation of [3]. The [4] of the Chinese Expert Consensus and Path Management Guide for Accelerated Rehabilitation Surgery (2018 edition) advocates the early postoperative recovery of diet. Studies have shown that the early recovery of oral eating, drinking water and early oral assisted nutrition after elective abdominal surgery can promote the recovery of intestinal motor function, help to maintain intestinal mucosa function, prevent microflora imbalance and displacement, and can reduce the incidence of postoperative infection and shorten the postoperative hospitalization time by [5]. At present, shortening the perioperative water fasting time needs to be concentrated in the preoperative stage. Although the guidelines and a small number of studies recommend the early recovery of diet after surgery, there is no clear stipulation on the recovery time of postoperative diet and drinking water, and most domestic hospitals still perform fasting for at least 6h after surgery.

Carbohydrates are perioperative good oral nutritional fluids. In recent years, studies have shown that preoperative oral carbohydrates can not only supplement the lost water and energy, improve their thirst and hunger, but also improve the postoperative metabolism and stress changes, reduce postoperative insulin resistance, shorten the hospital stay, and accelerate the <sup>[6]</sup> recovery of patients compared with clear water. Furthermore, preoperative oral carbohydrate has been confirmed by many studies and does not increase the risk of reflux aspiration in <sup>[7]</sup>. However, most of the current clinical studies of oral carbohydrate effects on postoperative recovery focus on the preoperative oral phase, and only a few small samples have shown that postoperative oral carbohydrate improves postoperative comfort <sup>[8]</sup>. Therefore, further systematic studies on the effects of early postoperative oral carbohydrates on postoperative recovery remain lacking.

## **Directory of reference**

[1] Miller TE, Roche AM, Mythen M. Fluid management and goal-directed therapy as an adjunct to Enhanced Recovery After Surgery (ERAS). Can J Anaesth. 2015 Feb;62(2):158-68.

- [2] Rizvanović N, Nesek Adam V, Čaušević S, Dervišević S, Delibegović S. A randomised controlled study of preoperative oral carbohydrate loading versus fasting in patients undergoing colorectal surgery. Int J Colorectal Dis. 2019 Sep;34(9):1551-1561. doi: 10.1007/s00384-019-03349-4. Epub 2019 Jul 15. PMID: 31309323.
- [3] Nygren J, Thorell A, Ljungqvist O. Preoperative oral carbohydrate therapy. Curr Opin Anaesthesiol. 2015 Jun;28(3):364-9. doi: 10.1097/ACO.0000000000000192. PMID: 25827282.
- [4] Surgery Branch of Chinese Medical Association, Anesthesiology Branch of Chinese Medical Society. Chinese Expert Consensus and Path Management Guidelines for Accelerating Rehabilitation Surgery (2018) [J]. Chinese Journal of Anesthesiology, 2018,38 (001): 8-13.
- [5] Yang R, Tao W, Chen YY, Zhang BH, Tang JM, Zhong S, Chen XX. Enhanced recovery after surgery programs versus traditional perioperative care in laparoscopic hepatectomy: A meta-analysis. Int J Surg. 2016 Dec;36(Pt A):274-282. doi: 10.1016/j.ijsu.2016.11.017. Epub 2016 Nov 10. PMID: 27840308.
- [6] Bethune Orthopaedic Accelerated Rehabilitation Alliance, Bethune Charity Foundation Orthopaedic Professional Committee of trauma, Joint Surgery Professional Committee of Bethune Charity Foundation, etc. Guidelines for the management of perioperative fasting fasting in orthopaedic surgery [J]. Chinese Journal of Trauma and Orthopedics, 2019,21 (10): 829-834.
- [7] MD Smith, Mccall J, Plank L, et al. Preoperative carbohydrate treatment for enhancing recovery after elective surgery[J]. Cochrane Database Syst Rev, 2014, 8(8):CD009161.
- [8] Noba L , Wakefield A . Are carbohydrate drinks more effective than preoperative fasting: A systematic review of randomised controlled trials[J]. Journal of Clinical Nursing, 2019, 28.
- [9] Wang Cuilan, Huang Yuting, Zeng Qing, et al. Study on postoperative fasting water prohibition time under ERAS concept [J]. Clinical Medical Engineering, 2022,29 (4): 2.

## 1. Study purpose and study endpoint

## 1.1 Study Purpose

- **1.1.1 Main study objective**: To evaluate the effect of oral carbohydrates early after TKA on the nutritional status of elderly patients.
- 1.1.2 Secondary study objectives: To evaluate the effect of early oral carbohydrate administration on the comfort and safety of TKA in elderly patients.
- 1.2 Study endpoint
- 1.2.1 Primary study endpoints

Pre-albumin levels in venous blood in the fasting state on the day of surgery, 1d and 3d after surgery.

- 1.2.2 Secondary study endpoints
- 1.2.2.1, Effectiveness study endpoint
- 1) The level of retinol-binding protein in venous blood on the day and 1d and 3d after surgery;
- 2) The insulin resistance index in venous blood was checked on the empty stomach on the morning, 1d and 3d after the operation;
- 3) NRS score of thirst and hunger at 2h, 6h and 8h after surgery;
- 4) Abating distension within 24h after surgery;
- 5) The incidence of hypoxemia and reflux aspiration within 24h after surgery;
- 6) Time of anal exhaust for the first time after surgery;
- 7) Time to leave bed for the first time after surgery;
- 8) Length of hospitalization;
- 9) Postoperative subject satisfaction score.
- 1.2.2.2. Safety study endpoint
- 1) The incidence and severity of various adverse events (AE) from the start of oral carbohydrates to the end of the trial;
- 2) The incidence and severity of adverse events such as nausea, vomiting and hypoxemia from the first start of drug administration to the end of the trial;
- 3) Number of antiemetic drugs used within 24h after the first start to the first start of drug administration;
- 2. Expected results

Oral carbohydrates in the early postoperative period can improve patient nutritional

status, improve comfort and satisfaction without increasing the incidence of adverse events.

## 3. Design and method of the study

## 3.1.1 Screening period

Patients with elective knee replacement, screened with informed consent to enroll patients, met all enrollment criteria and did not meet any of the exclusion criteria.

#### 3.1.2 Treatment Period

Actively control blood pressure, blood pressure and blood sugar, correct anaemia and hypoproteinemia, and increase protein intake before surgery. The dietary plan was informed by the ward nurse: all patients were fasted with solid food 6 hours before surgery and took 200 milliliters of carbohydrates orally 2-3 hours before surgery.

The venous access was open after home invasion and was routinely monitored electrocardiogram(ECG), non-invasive blood pressure(NBP), oxygen saturation(SpO2), bispectral index (BIS). Parecoxib 40 milligrams of analgesia was given intravenously at 30 minutes before the start of the procedure. Adductor canal block (ACB) and Infiltration between poplitealartery and capsule of knee (IPACK) block were performed on the lower limbs of the surgical side using an ultrasound high-frequency line array probe before induction of the general anesthesia procedure.

Anesthesia induction: after static injection of Midazolam 0.03 milligrams / kilogram, Propofol 2 milligrams / kilogram, Sufentanyl 0.4 milligrams / kilogram, Cisatracurium 0.2 milligrams / kilogram. The tracheal tube was inserted after 3minutes and mechanical controlled ventilation was performed mechanical controlled ventilation, fraction of inspired oxygen (FiO2) 40%, oxygen flow 2 litres/ minutes, minute ventilation 7 milliliters / kilogram, respiratory rate (RR) 12 times/ inspiration-to-expiratory ratio (I: E) 1:2, maintain partial pressure of carbon dioxide in endexpiratory gas (PETCO2) 35-40 millimeters of mercury (mmHg). Anesthesia maintenance: intravenous propofol 4~7 milligrams / kilogram/ hour, remifentanl 0.3-0.5 microgrammes/kilogram/ hour, maintain BIS 40~60. A restrictive fluid management strategy was adopted, with 6ml/ kg·h supplemented with physiological needs, blood loss was supplemented with hydroxyethylstarch fluid, and concentrated red blood cells were infused at hemoglobin (Hb) <80 grams / litre to maintain patient blood pressure and heart rate fluctuations less than  $\pm 20\%$  of the basal value . Dexamethasone 5mg and totoxetron 2mg for prophylactic antiemesis were given intravenously at 30min before the end of the surgery. All patients used hydromorphone patient-controlled intravenous analgesia (PCIA) continuous: 1ml / h, automatic control: 5ml, locking: 10min, limit: 35ml / h, adjust parameters according to the pain.

Internal postanesthesia care unit (PACU) management: Patients will randomly enter

the PACU into two study groups: early carbohydrate feeding group (EOF group) and conventional feeding group (control group). Routine feeding group (Group C): Patients in group C were observed with 60min of abnormal vital signs after extubation, and returned to the ward for fasting and fasting for at least 6 h, and began to eat gradually through the mouth after anal exhaust. Early carbohydrate feeding group (EOF group): The EOF group drank 10.5% of 5 ml/kg body weight (100ml containing 12.5g maltodextrin, fructose and glucose) after extubation in the resuscitation room. PACU management: Patients will randomly enter the PACU into two study groups: early carbohydrate feeding group (EOF group) and conventional feeding group (control group). Routine feeding group (Group C): Patients in group C were observed with 60min of abnormal vital signs after extubation, and returned to the ward for fasting and fasting for at least 6 h, and began to eat gradually through the mouth after anal exhaust. Early carbohydrate feeding group (EOF group): The EOF group drank 10.5% of 5 ml/kg body weight (100ml containing 12.5g maltodextrin, fructose and glucose) after extubation in the resuscitation room.

To evaluate the drinking criteria for patients in the EOF group: Steward wake score of 6 and wake level level 3, take 5 ml/kg body weight of 12.5% carbohydrate (100ml containing 12.5g maltodextrin, fructose, and glucose) according to the patient's consent. The process of drinking carbohydrates was to take 30ml orally first. After observing the swallowing without abnormality, the patient was ordered to drink the remaining drinks within 2h. After the patient returned to the ward, the liquid diet began to gradually overenter the normal diet. When the patient was able to tolerate the normal diet, v.

Evaluation process of the drinking index:

- 1. Steward score: Akefulness: 0-no response to stimulus; 1-some response to stimulus; 2-full awake.(2) Respiratory tract patency degree: 0 points-the patient's respiratory tract needs support; 1 points-the patient's respiratory tract can maintain patency without support; 2 points-the patient can cough according to the doctor's guidance.(3) Body activity degree: 1 points-the patient's limb has no activity; 2 points-the patient's limb has an unconscious activity; 3 points-the patient's limb can carry out conscious activities
- 2. Wakefulness classification according to the patient's consciousness performance: Level 0: the patient is completely asleep, Call without any response; Level 1: The patient is falling asleep, However, head and neck movement, eye opening or limb movement when breathing; level 2: the patient is awake, Have the same performance as level 1, At the same time can also open the mouth, stretch the tongue; Level 3: The patient is awake, Have the same performance as level 2, At the same time can also clearly say their own name, age and other information; Level 4: The patient is awake, Have the same performance as level 3, It can also accurately identify the surrounding environment, And tell you exactly where you are.
- 3. In addition to receiving different feeding treatment programs in the PACU, the two groups received the same care and diet program formulated by the same care group.
- 3.1.3 The Follow-up Period

Record: Patients had fasting serum prealbumin, retinol-binding protein levels, and

insulin resistance index on the same day, 1day and 3 days after surgery.

Record: 2 hours, 6 hours and 8 hours postoperative digital scores; bloating, hypoxemia and reflux aspiration occurred 24 hours after surgery.

Record: length of hospitalization, first anal exhaust time, first ambulation time, nausea and vomiting, and patient satisfaction.

- 4. Subject recruitment and protective measures
- 4.1 Inclusion criteria
- Patients undergoing elective knee replacement surgery;
- the patient gave informed consent;
- Age  $\geq$ 65 years, Sex is not limited
- American Society of Anesthesiologists(ASA)I~III level
- Body Mass Index(BMI)18~28kg/m2
- 4.2 Exclusion criteria
- Preoperative gastric emptying disorders, such as gastroesophageal reflux or previous surgery;
- Diabetes mellitus, severe renal insufficiency, or other severe metabolic diseases;
- History of motion sickness;
- Mental disorders, alcoholism, or a history of substance abuse;
- Patients with abnormal swallowing function;
- Maltodextrin, fructose allergy or intolerance;
- Surgery time was greater than 3 hours.

#### 4.3 Exit criteria

Patients may withdraw their informed consent and withdraw from the trial at any time.

The investigator may decide on the subject to terminate the withdrawal from the study in the following circumstances.

Any medical condition in the study leads to the risk of continuing the study subjects; Subjects receive analgesic treatment other than the prescribed analgesic remedy protocol, and other subjects who fail to complete the test as specified in the test protocol;

The investigator judged the other conditions that should be withdrawn from the trial.

5 Informed consent

#### 5.1 The Informed Consent Form

The informed consent was in accordance with the ethical principles outlined in the Declaration of Helsinki. The informed consent form detailed the study protocol and process, and fully explained the risks of the study.

The informed consent form also states that the records of the individual identity must be kept confidential, but the research team and regulators can access the subject information.

## 5.2 Informed consent process and record

Informed consent begins before the individual consent to participate in clinical studies and continued throughout the course of the clinical study.

#### 5.3 Confidential

Personal patient information will be given as confidential information. All patient data

obtained from the patient cases will be kept as confidential. Patients will be identified by their name acronym and the numbers provided at the time of study inclusion. Patients or their families will be aware of the anonymity of the data and their right to protect their privacy. However, it is also important to understand the fact that the data will be submitted to the subject responsible unit or the government management authority, and may also be submitted to institutions such as the Ministry of Health for inspection and evaluation. The participating physician will keep a list of patient personal data (patient data and corresponding patient names) for confirmation of the record.

#### 6. Quality control and quality assurance

## 6.1 Qualification of research unit and researcher qualification

The research unit shall have the experience in drug research, the facilities and conditions of the department where the project belongs shall meet the needs of safe and effective clinical research, and the researchers shall have the professional expertise, qualifications and ability to undertake the clinical research, and shall be trained in GCP regulations.

## 6.2 Training of the researchers

Before the start of the study, the research leaders of each center should organize the researchers to study the program, and only the researchers who have passed the program training can participate in the study to ensure that the researchers have a consistent understanding of the protocol. For important assessment scales, relevant personnel in the participating centers need systematic training and even obtain corresponding qualification certificates.

## 6.3 Surveillance of clinical trials

The hospital ethics committee and institutional review board may conduct a systematic review of the clinical trial-related activities and documents, to evaluate whether the trial was conducted in accordance with the test protocol, SOP, and relevant regulations, and whether the test data are timely, true, accurate, and complete records. The audit should be performed by those who do not directly involve the clinical trial.

## 7. Organization and management of the research

## 7.1 Change of the scheme

All additional or referenced appendices are integral parts of the scheme. No one shall make any modifications or revisions to any part of the research protocol, as signed by the investigator and the principal of the project, unless these changes or revisions have been fully discussed. And through the unanimous consent of the researcher and the subject leader.

Any agreed modifications will be recorded and will be signed by the investigator and the project leader and filed with the protocol.

## 7.2 Retention of the records

The investigator shall keep all the detailed original documents of the subject and record the trial process, medication status, laboratory examination data, safety data and efficacy assessment in the case report form. The recorded data shall be complete, timely and clear. The original documents and medical records should be clear, detailed

and easily identified by those participating in this clinical trial.

The case report form and the original files can only be modified by the investigator. No modification to the case report form and the original file shall smear the original data off. The correct way to modify is to line the original data, and then write the modified data next to the original data, and sign the date and the name of the modification.

Test data shall be retained until 5 years after the termination of the test.

## 7.3 Early termination of the study

The leader of the project decides to stop or interrupt the study in advance in the case of force majeure, and should inform the doctors involved in the study in writing. Similarly, any participating unit that decides to withdraw from the study for any reason should also notify the project leader in written form.

7.4 Research, supervision and inspection

## 7.4.1 Research supervision

Inspectors must follow the drug clinical trial quality management specification (GCP) and standard operation procedures (SOP), visit the research unit regularly or according to the actual situation, supervise the clinical trial work and progress, check, confirm all data records and reports, correct and complete, consistent with the original data, ensure the clinical trial in accordance with the clinical trial protocol, the researchers should actively cooperate with the inspectors. The specific contents of the inspector include:

- a) Ensure that the test undertaking unit has appropriate conditions, including staffing and training, complete laboratory equipment, good operation, various inspection conditions related to the test, an estimated sufficient number of subjects, and the participants to be familiar with the requirements in the test plan;
- b) Monitor the implementation of the trial program during the trial, confirm that the informed consent of all subjects is obtained before the trial, understand the enrollment rate of the subjects and the progress of the trial, and confirm that the selected subjects are qualified;
- c) Confirm that the records and reports of all data are correct and complete, and that all case report forms are entered correctly and consistent with the original data. All errors or omissions have been corrected or indicated, signed and dated by the Investigator.
- d) Verify that all adverse events are recorded, and that serious adverse events shall be reported and recorded within the specified time;
- e) Clearly and truthfully record the failed visits, unconducted tests, and undone checks should be made, and whether the errors and omissions should be corrected;
- f) The written inspection report shall be completed after each visit, which shall state the date, time, name of the inspector, the findings of the inspection, etc.

## 7.4.2 On-site inspection

The responsible unit may conduct an on-site inspection of the research at a clinical research institution. The audit includes the required test documents, records of the informed consent process, and the consistency of the eCRF and the original documents. But also the content and scope of the inspection can be increased

according to the situation. The investigator agrees to participate at a reasonable time and in a reasonable manner.

8. Investigators' responsibilities

## 8.1 Participation of doctor responsibilities

The participating physicians will conduct the study following the study protocol and confirm the accuracy of the data entered. The participating physicians should be responsible for obtaining written signed informed consent for data collection from the study subjects.

## 8.2 Responsibility of the project leader

The project leader takes all reasonable steps and provides sufficient resources to ensure the implementation of the research, mainly involving the following aspects:

- a) Ensure that the study complies with relevant national and local regulations, including ethical requirements, patient data protection regulations, etc.
- b) Ensure the effectiveness of quality control and analysis of research results.
- 9. Share results

The intellectual property rights, trial data and research results related to this study are jointly owned by Nanjing First Hospital and the Department of Anesthesiology.

The intellectual property rights, trial data and research results related to this clinical study are owned by Nanjing First Hospital and the Anesthesiology Department.

10. Ethics principles and requirements for clinical research

Clinical research will follow the world medical congress "declaration of Helsinki" and the national health and family planning commission of the People's Republic of China "involving people biomedical research ethics review method" and other relevant provisions, the specific implementation of informed consent, the privacy protection, research free and compensation, risk control, special subject protection and research related damage compensation principles and requirements. The clinical study was performed before the ethics committee approved the trial protocol. Before each subject is enrolled in the study, the investigator has the responsibility to present the subject or / and his legal agent about the purpose, procedures of the study and possible risks, and sign a written informed consent form that their participation in the clinical study is completely voluntary, that they may refuse to participate or withdraw from the study at any time at any stage of the trial without discrimination and retaliation, and their medical treatment and interests are not affected. The informed consent form should be retained as a clinical research document for future reference to effectively protect the subjects' personal privacy and data confidentiality.